CLINICAL TRIAL: NCT02845726
Title: Biofilms on Short-term Indwelling Ureteral Stents: Influence on Associated Symptoms and Complications; Prediction by Urine Analysis; Current Bacterial Spectrum and Antibiotic Resistance
Brief Title: Biofilms on Short-term Indwelling Ureteral Stents
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Dominik Abt, Dr. med., Cantonal Hospital of St. Gallen
Other Study IDs: CTU 15.010
Record Dates: First submitted 2016-07-08; First posted 2016-07-27 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Ureteral Catheterization; Biofilm; Morbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with temporary ureteral stent: Assessment of patients transiently undergoing ureteral stenting.
  Interventions: Other: Stent examination, urinary analysis, USSQ questionnaire

INTERVENTIONS:
Other: Stent examination, urinary analysis, USSQ questionnaire

SUMMARY:
This study is performed to analyze various aspects of biofilms on ureteral stents.

DETAILED DESCRIPTION:
The study is performed to provide a better understanding of the influence of biofilms on ureteral stents on the entire spectrum of stent-associated morbidity.

Moreover, it could provide more detailed knowledge about the correlation of the occurrence of biofilms on ureteral stents and findings in urinary analysis, which could serve as a decision support whether patients with ureteral stents undergoing further interventions (for example ESWL or simple secondary URS) should receive antibiotic prophylaxis.

Correlation of results of urinary bacteriologies (assessed pre- and intraoperatively) and biofilm analysis on stents could provide information if "targeted antibiotic treatment" based on urinary bacteriology only is possible at all.

Correlation of urinary analysis and conventional urinary bacteriology could provide a valuable contribution regarding the prediction of bacteriuria and the necessity of postponing operations.

Additionally, the study is intended to provide an overview over the recent bacterial species that are involved into biofilms on ureteral stents and their resistance to antibiotics. This could provide valuable information about the choice of antibiotics in cases were treatment has to be performed empirically.

ELIGIBILITY:
Inclusion Criteria:

* Patients temporarily undergoing ureteral stenting
* Informed consent

Exclusion Criteria:

* Bilateral stenting
* Ureteral obstruction due to malignancies
* Additionally performed procedures/operations during stent indwelling time -Cognitively impaired patients
* UTI at the time of stent insertion (>10 to the power of 2 cfu/ml)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing ureteral stenting for the preparation of a secondary intervention in an inpatient setting at the department of urology of KSSG.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-09-23 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Total biofilm mass on ureteral stents. | Time of stent removal: Four weeks (range 2-6 weeks) after stent insertion
Assessment of morbidity using the Ureteral Stent Symptom Questionnaire (USSQ) | Day before stent removal (i.e. 4 weeks (range 2-6 weeks) after insertion)

SECONDARY OUTCOMES:
Assessment of morbidity using the Ureteral Stent Symptom Questionnaire (USSQ) | One week after stent insertion; Four weeks (range 2-6 weeks) after stent removal.
Urinary analysis (pH, nitrite, leucocyturia, hematuria). | Day before stent removal (i.e. 4 weeks (range 2-6 weeks) after insertion)
Urine Culture | Before study inclusion; Day before stent removal (i.e. 4 weeks (range 2-6 weeks) after insertion); Intraoperatively (during stent removal)
Rapid immunoassay test for bacteriuria | Day before stent removal (i.e. 4 weeks (range 2-6 weeks) after insertion)
Next generation sequencing of biofilms | Day of stent removal: Four weeks (range 2-6 weeks) after stent insertion
  To identify bacterial species that are involved into biofilms on ureteral stents.
Number of bacteria on stent surface (cell count as estimated by scanning electron microscopy) | Day of stent removal: Four weeks (range 2-6 weeks) after stent insertion
Number of bacteria on stent surface (determined via quantitative PCR) | Day of stent removal: Four weeks (range 2-6 weeks) after stent insertion

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Abt, Dr. med., Principal Investigator — Department of Urology
Locations (1):
- Urological Department, Cantonal Hospital of St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buhmann MT, Abt D, Nolte O, Neu TR, Strempel S, Albrich WC, Betschart P, Zumstein V, Neels A, Maniura-Weber K, Ren Q. Encrustations on ureteral stents from patients without urinary tract infection reveal distinct urotypes and a low bacterial load. Microbiome. 2019 Apr 13;7(1):60. doi: 10.1186/s40168-019-0674-x. PMID 30981280